CLINICAL TRIAL: NCT03812211
Title: Evaluation of a Supplement for Weight Management in Obese and Overweight Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Principal Investigator, Mark Tarnopolsky, Principal Investigator, Professor, Director of Neuromuscular and Neurometabolic Clinic, McMaster University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 5754
Record Dates: First submitted 2019-01-18; First posted 2019-01-23 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Overweight and Obesity; Men; Women
MeSH Terms: conditions — Overweight; Obesity; Multiple Endocrine Neoplasia Type 1

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Supplement (Active Comparator): Participants will be allocated in a randomized, double-masked manner to receive a multi-faceted supplement for the 12-week duration of the study
  Interventions: Dietary Supplement: Active Supplement
- Placebo (Placebo Comparator): Participants will be allocated in a randomized, double-masked manner to receive a placebo supplement (the placebo will be made of microcrystalline cellulose, and will be matched in size, appearance, taste and caloric value) for the 12-week duration of the study
  Interventions: Dietary Supplement: Placebo supplement

INTERVENTIONS:
Dietary Supplement: Active Supplement — Examine the effects of a multi-faceted supplement comprised of vitamins, minerals and naturally occurring and plant extracts approved for consumption of in overweight/obese men and women
  Arms: Active Supplement
Dietary Supplement: Placebo supplement — Examine the effects of a placebo supplement in overweight/obese men and women, compare to the active supplement
  Arms: Placebo

SUMMARY:
The purpose of this trial is to examine the effects of a novel, orally consumed dietary supplement (composed of naturally occurring components) on weight management and metabolic rate in individuals who are overweight or obese following a 12-week supplementation period. The investigator's primary outcome will be changes in body composition measured via dual energy x-ray absorptiometry (DXA), which will measure changes in fat and lean mass during the supplementation period. Another primary objective will be to determine whether or not the body mass index (BMI) changes during the supplementation period. A secondary objective of the study is to determine whether anthropometric measurements (waist-to-hip ratio) is altered following the supplementation period. Another secondary objective of this study is to determine whether metabolic rate (as measured in VO2 consumption at rest and during exercise) is changed following the supplementation period. Another secondary objective is to determine whether blood pressure (systolic and diastolic pressure, measured in mm Hg) and physical function (measured via VO2peak in mL/min/kg-1 and leg strength in kilograms) change when the supplement is administered over a 12-week period. Another secondary objective will determine how glycemic control, blood markers of inflammation and cholesterol are affected by this intervention.

DETAILED DESCRIPTION:
The present study is a randomized double-blind placebo controlled repeated measures design, with sampling of the cohorts on five separate occasions.

Group 1: Intervention Group (n = 24) Healthy, overweight or obese physically inactive males, supplement, n = 12 Healthy, overweight or obese physically inactive females, supplement, n=12 Group 2: Placebo Group (n = 24) Healthy, overweight or obese physically inactive males, no supplement, n = 12 Healthy, overweight or obese physically inactive females, no supplement, n=12

Participants will be asked to make 5 visits.

Day 0 (Visit 1): Eligible participants that provided informed consent will complete a medical screening questionnaire to determine their readiness to perform exercise. Participants will thus complete the SF-36 and CSEP Get Active Questionnaire form. Participant characteristics will then be measured. At this time, anthropometric measurements (i.e., height, weight, waist circumference) and a dual energy x-ray absorptiometry (DXA) measurement will be performed. This must be done in order to verify that the participant meets the inclusion criteria of being overweight. Following this screening, participants will begin the following the study timeline.Upon completion, participants will be randomized into one of two groups.

Day 1 (Visit 2): Participants will arrive following an overnight fast (including no caffeine for 12 hours) and having abstained from any exercise for the prior 48 hours. Participants will enter the clinic, and rest quietly in the supine position for 25 minutes before having blood pressure with a non-invasive automated cuff and resting metabolic rate via metabolic cart measured. Following resting blood pressure and baseline metabolic rate assessment, blood will be drawn from an antecubital vein. Thereafter, functional metrics will be determined including strength (both upper and lower body muscles; and aerobic capacity (V02peak). Following testing, participants will be provided with a 3-day diet log (which will be completed every two weeks) and a pedometer.

Day 14 (Visit 3); Participants will arrive following an overnight fast (including no caffeine for 12 hours) and having abstained from any exercise for the prior 24 hours. Participants will undergo a DXA. Blood will be drawn from an antecubital vein.

Day 49 (Visit 4); Participants will arrive following an overnight fast (including no caffeine for 12 hours) and having abstained from any exercise for the prior 24 hours. Participants will undergo a DXA.

Follow-up - Day 7, 21, 28, 35, 42, 56, 63, 70, 77: Participants will receive a weekly phone call to determine their pedometer counts for the week, and to ensure that participants are adhering to the supplement consumption, and to address any concerns.

Day 84 (Visit 5); Participants will repeat Day 1 (automated blood pressure, resting and maximal metabolic rate, blood draw, functional metrics. Participants will return their pedometer and remuneration will be processed.

Study products (active supplement vs. placebo) will be provided in a blinded fashion by Infinit Nutrition Canada (Windsor, Ontario). The active supplement is composed of vitamins, minerals and naturally occurring and plant extracts approved for consumption. Participants will be asked to consume 3 servings of the study product per day (7 days per week) throughout the 12-wk intervention period. Participants will consume 1 serving immediately before breakfast. Participants will be instructed to consume the supplement in a single sitting, with water, within 5-10 min. Participants will be instructed to record product intake in a diary to check compliance. Participants will also be asked to maintain the used package and turn it in at the check-ins as a marker of study compliance. To maintain the double-blind nature of the experiment, the placebo, which contains microcrystalline cellulose, will be matched in size, appearance, taste and caloric value

Three day weighed food record. Participants will be asked to record everything that they consumed for 3 non-consecutive days: 2 week-days and either a Saturday or a Sunday. On completion of the food record, it will be analyzed using a commercially available computerized database software (Nutribase version 11.5, Cybersoft Inc., Phoenix, AZ, USA). Food items will be aggregated into the following categories: fruit (e.g., fresh/frozen, tinned, juice), vegetables (e.g., fresh/frozen, canned), dairy products (e.g., milk, yoghurt, cheese), breads and cereals (e.g., bread, breakfast cereal, rice, pasta), meats and alternatives (e.g., red meat, poultry, fish, pork, processed meat, tofu, eggs, nuts) and extra foods (e.g., hamburger, pizza, meat pies, chocolate, cake, ice cream, jam, biscuits, crackers, crisps, alcohol etc.).

Resting metabolic rate (RMR). Participants will be asked to lay still on a bed will connected to a metabolic cart with an on-line gas collection system (Moxus modular oxygen uptake system, AEI Technologies, Pittsburgh, PA), and the system will acquire oxygen consumption (VO2) and carbon dioxide (CO2) production data for 15 minutes.

Blood sampling. A total of ~16 mL blood per visit will be taken from the antecubital vein and drawn into evacuated tubes with heparin used for plasma collection and non-treated tubes will be used to collect serum. Blood sampling will be used for the following panel of tests: complete blood count (CBC), glucose, Gamma-Glutamyl Transferase (GGT), bilirubin, Alanine Aminotransferase (ALT), creatine kinase (CK), creatinine, triglycerides, total cholesterol, LDL and HDL, insulin, CRP, and leptin.

Maximal voluntary VO2peak fitness test. Participants will complete double-leg incremental peak oxygen uptake (VO2peak) tests on a cycle ergometer (Lode, Groningen, the Netherlands). A metabolic cart with an on-line gas collection system (Moxus modular oxygen uptake system, AEI Technologies, Pittsburgh, PA) will acquire oxygen consumption (VO2) and carbon dioxide (CO2) production data. For double-leg cycling, the test will begin with a 1-min warm up at 50 watts (W), after which the power will be increased by 1 W every two seconds until volitional exhaustion or the point at which pedal cadence falls below 60 rpm. Heart rate will be monitored continuously throughout the test via telemetry with a heart rate monitor (Polar A3, Lake Success, NY). VO2peak will be defined as the highest oxygen consumption achieved over a 30-s period. Maximal workload (Wmax) will be the highest power output achieved during the test. After the completion of the test, the participant will be asked to perform a 2-3-minute active recovery pedaling against no resistance.

Pedometer. Participants will be given a wearable activity tracker (pedometer). All participants will record their daily totals for subsequent analysis.

Dual X-ray absorptiometry (DXA) and blood pressure. A DXA scan is a non-invasive procedure requiring the participant to only lay still on a padded table. It is a fast procedure that provides a variety of body composition variables (bone mass/area/density, fat mass, and fat free mass). The DXA scan exposes individuals to low levels of radiation, approximately 0.18 millirem. According to the United States Nuclear Regulatory Commission, Americans receive approximately 620 millirem each year, half of which is due to environmental background radiation. Radiation exposure can be due to medical treatments or procedures, like X-Ray or MRI's, food, sun exposure, etc. Any exposure to radiation can increase the risk of cancer. In the present study, body composition will be assessed using DXA scan (GE Lunar Prodigy, Madison, WI) and a software program for adults (encore Version 9.15.010). Fat free mass (FFM), fat mass (FM) and bone mineral density (BMD) of the entire body will be recorded. Arterial blood pressure (i.e., systolic [SBP] and diastolic [DBP]) will be measured during rest with a stethoscope (Marshall Nurse Stethoscope, Riverside, Ill., USA) and sphygmomanometer (MDF Instruments Direct Inc., Agoura Hills, Calif., USA).

Waist and hip circumference measures. For waist circumference measurement, the participant will stand with arms at the sides, feet together, and abdomen relaxed. Using a Gulick tape measure, a horizontal measure will be taken at the narrowest part of the torso (above the umbilicus and below the xiphoid process). Obtaining a horizontal measure directly above the iliac crest enhances standardization according to The National Obesity Task Force. For hip circumference measurement, the participant stands erect and feet together, a horizontal measure is taken at the maximal circumference of buttocks.

Leg press 1RM. Assessment procedures for determining lower body strength using leg press exercise equipment (Cybex Eagle ®, Medway, MA) will require the participant to sit in the leg press machine with the right foot and left foot on the weight platform. The seat and back pad will be adjusted so that feet are flat on the platform hip-width apart, toes slightly angled out, and legs parallel to each other. The interviewer will then instruct the participant to grasp the handles or sides of the seat and extend their legs leaving just a slight bend in the knee. Next, the participant will remove the racking mechanism from the platform and grasp the handles or seat again. The participant will begin with a selected weight that is within their perceived ability, approximately 60 to 80% of maximum capacity (make an educated guess). The participant will lower the platform slowly and controlled towards the chest, keeping the hips and buttocks on the seat, and the back flat against the back pad. Once the thighs are parallel to the platform the participant will extend the legs, pushing the weight back to the start position as hard and as fast as possible. The participant will be instructed to not allow their hips to shift to one side, the buttocks to rise, or knees to move inward or outward during this exercise. The interviewer will also instruct the participant to keep heels flat and not allow the knees to go beyond the toes. Once the repetitions are completed, the participant will replace the racking mechanism and exit the leg press. These procedures were adapted from procedures described by the National Strength and Condition Association (2008) and the American College of Sports Medicine (2013).

Hand grip strength (MVIC; maximum voluntary isometric contraction). Hand grip strength will be measured using an isometric dynamometer (JAMAR®, Sammons, Bolingbrook, IL). The grip width will be adjusted to hand size and with arm flexed at 90°, the participant will perform three X 5 s efforts with a one min rest between trials.

Knee extension (MVIC;maximum voluntary isometric contraction). Isometric knee extension will be measured by mechanical dynamometry (Biodex System 3, Biodex Medical Systems, Shirley, NY). Participants will be positioned into the machine with the knee flexed at 90° and perform three X 5s maximal voluntary contractions with 30s rest between each trial.

Questionnaires. The RAND 36-Item Health Survey (Version 1.0) taps eight health concepts: physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue, and general health perceptions. It also includes a single item that provides an indication of perceived change in health. The Get Active Questionnaire by CSEP is a 2-page, self-administered, pre-participation for exercise screening tool. Potential participants must answer 'no' to all questions on the Get Active Questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* overweight (BMI 25 - 29.9 kg/m2) or obese (BMI > 30 kg/m2)
* Physically inactive (< 1 hour of formal exercise/week)

Exclusion Criteria:

Participants will be excluded and/or released from the study if they meet any one of the following:

* Smoking
* Use of assistive walking devices (e.g., cane, or walker)
* Chronic use of analgesic or anti-inflammatory drugs
* Diabetes mellitus (more than one anti-diabetic drug)
* Cardiovascular disease (recent myocardial infarction (< 6 months) and/or hypertension requiring more than 2 medications)
* Congestive heart failure requiring more than one medication for control
* Renal disease (creatinine > 140)
* Previous stroke
* Active musculoskeletal injuries and/or severe osteoarthritis
* Significant weight loss in the 3-month period prior to the study
* Vegan diet
* Muscular dystrophy
* Severe peripheral neuropathy
* Severe osteoporosis
* Use medications known to affect protein metabolism (i.e. corticosteroids)
* Inability to consent
* Chronic obstructive pulmonary disease, and asthma requiring more than two medications.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 65 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-04-24 (Actual); Study Completion 2022-12-02 (Actual)

PRIMARY OUTCOMES:
Body composition | 12 weeks
  Fat free mass and fat mass measured via DXA
Body mass index | 12 weeks
  Measure of body fat based on height and weight that applies to adult men and women

SECONDARY OUTCOMES:
Blood pressure | 12 weeks
  systolic and diastolic pressure, measured in mm Hg
Muscle strength | 12 weeks
  Leg strength measured via Biodex
Aerobic fitness | 12 weeks
  VO2peak in mL/min/kg-1
Fuel source utilization | 12 weeks
  Consumed O2 compared to expired CO2
Hemaglobin A1C in mmol/mol | 12 weeks
  Amount of glycated hemoglobin
Concentration of insulin in the blood | 12 weeks
  Measures the amount of insulin in the blood.
Concentration of lipids in the blood | 12 weeks
  Cholesterol, low density lipoprotein, high density lipoprotein, triglycerides in the blood
Quality of Life rating | 12 weeks
  RAND SF(short form health survey)-36 Questionnaire; The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability
Anthropometric measurements | 12 weeks
  Waist-to-hip ratio measurements (in cm)

CONTACTS AND LOCATIONS:
Locations (1):
- McMaster University Medical Center, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Godard MP, Johnson BA, Richmond SR. Body composition and hormonal adaptations associated with forskolin consumption in overweight and obese men. Obes Res. 2005 Aug;13(8):1335-43. doi: 10.1038/oby.2005.162. PMID 16129715
- [Background] Bailey SJ, Winyard P, Vanhatalo A, Blackwell JR, Dimenna FJ, Wilkerson DP, Tarr J, Benjamin N, Jones AM. Dietary nitrate supplementation reduces the O2 cost of low-intensity exercise and enhances tolerance to high-intensity exercise in humans. J Appl Physiol (1985). 2009 Oct;107(4):1144-55. doi: 10.1152/japplphysiol.00722.2009. Epub 2009 Aug 6. PMID 19661447
- [Background] Cordero MD, Cano-Garcia FJ, Alcocer-Gomez E, De Miguel M, Sanchez-Alcazar JA. Oxidative stress correlates with headache symptoms in fibromyalgia: coenzyme Q(1)(0) effect on clinical improvement. PLoS One. 2012;7(4):e35677. doi: 10.1371/journal.pone.0035677. Epub 2012 Apr 19. PMID 22532869
- [Background] Maki KC, Reeves MS, Farmer M, Yasunaga K, Matsuo N, Katsuragi Y, Komikado M, Tokimitsu I, Wilder D, Jones F, Blumberg JB, Cartwright Y. Green tea catechin consumption enhances exercise-induced abdominal fat loss in overweight and obese adults. J Nutr. 2009 Feb;139(2):264-70. doi: 10.3945/jn.108.098293. Epub 2008 Dec 11. PMID 19074207
- [Background] Rasool AH, Yuen KH, Yusoff K, Wong AR, Rahman AR. Dose dependent elevation of plasma tocotrienol levels and its effect on arterial compliance, plasma total antioxidant status, and lipid profile in healthy humans supplemented with tocotrienol rich vitamin E. J Nutr Sci Vitaminol (Tokyo). 2006 Dec;52(6):473-8. doi: 10.3177/jnsv.52.473. PMID 17330512
- [Background] Thom E. The effect of chlorogenic acid enriched coffee on glucose absorption in healthy volunteers and its effect on body mass when used long-term in overweight and obese people. J Int Med Res. 2007 Nov-Dec;35(6):900-8. doi: 10.1177/147323000703500620. PMID 18035001
- [Background] Zembron-Lacny A, Slowinska-Lisowska M, Szygula Z, Witkowski K, Stefaniak T, Dziubek W. Assessment of the antioxidant effectiveness of alpha-lipoic acid in healthy men exposed to muscle-damaging exercise. J Physiol Pharmacol. 2009 Jun;60(2):139-43. PMID 19617657